CLINICAL TRIAL: NCT05247242
Title: Physical Activity and Social Engagement Program for Persons With Disabilities and Chronic Health Conditions in an Underserved Birmingham Community
Brief Title: Physical Activity and Social Engagement for Persons With Disabilities in an Underserved Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Lakeshore Foundation (Other)
Responsible Party: Principal Investigator, Laurie A Malone, PhD, Researcher IV, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB - 300008762; IRB-300008762 (Other: Center for the Study of Community Health, UAB)
Record Dates: First submitted 2022-01-18; First posted 2022-02-18 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Disability Physical; Chronic Conditions, Multiple; Aging
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tarrant Community Fitness Program: LOF-VR (Experimental): LOF-VR
  Interventions: Behavioral: Lakeshore Online Fitness (Online); Behavioral: Get Active with Virtual Reality (VR)
- Tarrant Community Fitness Program: VR-LOF (Experimental): VR-LOF
  Interventions: Behavioral: Lakeshore Online Fitness (Online); Behavioral: Get Active with Virtual Reality (VR)

INTERVENTIONS:
Behavioral: Lakeshore Online Fitness (Online) — Online physical activity program delivered to residents of Tarrant, AL via teleconferencing technology to a local community center. Instructors from Lakeshore will lead the physical activity program. This intervention will last six weeks.
Behavioral: Get Active with Virtual Reality (VR) — Participants will utilize the Oculus Quest 2 virtual reality headset, which is a head-mounted display system where users can interact with a virtual environment in a gaming setting. The Oculus Quest 2 incorporates social features where participants can interact with other users. This VR intervention will include periods of gameplay where participants can play games in either competitive or cooperative settings. This intervention will last six weeks.

SUMMARY:
Using a community-based participatory approach, this project aims to evaluate the feasibility, acceptability, and preliminary efficacy of two technology-driven group activity programs on socioemotional health and physical activity in a local underserved community, Tarrant, Alabama. Participants will complete two six-week programs, specifically Lakeshore Online Fitness (Online) and Get Active with Virtual Reality (VR).

DETAILED DESCRIPTION:
This project will utilize a cross-over randomized design where participants will initially be randomized into either the Online or VR intervention group. After completing the initial six weeks of the assigned intervention, participants will cross over and complete six weeks of the other intervention. No washout period is included due to several reasons, including no known washout period for certain socioemotional outcomes have been established by prior literature, ethical concerns in requiring return to baseline levels during washout, and a prolonged washout period would negatively impact participant adherence and retention to the study. Psychosocial metrics will be collected at the end of each activity session through surveys.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Tarrant, Alabama
* 18 years or older with a physical disability or chronic health condition or older than 60 years
* Fluent in English

Exclusion Criteria:

* Visual impairment that interferes with television viewing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Change in Social Isolation from Baseline to 12 weeks | 12 Weeks
  PROMIS Item Bank v2.0 - Social Isolation - SF 8a

SECONDARY OUTCOMES:
Change in Self-efficacy from Baseline to 12 weeks | 12 Weeks
  Self-efficacy for Exercise (SEE) Scale
Change in Loneliness from Baseline to 12 weeks | 12 Weeks
  NIH Toolbox Item Bank v2.0-Loneliness (Ages 18+)-Fixed Form
Change in Positive Affect from Baseline to 12 weeks | 12 Weeks
  NIH Toolbox Item Bank v2.0-Positive Affect
Change in Health-related quality of life from Baseline to 12 weeks | 12 Weeks
  SF-36v2
Change in Physical activity from Baseline to 12 weeks | 12 Weeks
  Physical Activity Scale for Individuals with Physical Disabilities (PASIPD)
Change in Enjoyment from Baseline to 12 weeks | 12 Weeks
  Visual Analog Scale (VAS) & Modified Physical Activity Enjoyment Scale (PACES)
Change in Physical Function from Baseline to 12 weeks | 12 Weeks
  Physical Function - Short Form 20a

CONTACTS AND LOCATIONS:
Locations (1):
- Tarrant Parks and Recreation, Tarrant, Alabama, United States

IPD SHARING:
Plan to Share IPD: No